CLINICAL TRIAL: NCT02961959
Title: Sacro-iliac Joint Arthrodesis or Non-operative Care for Treatment of Chronic Pelvic Pain. A Randomized Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spinal Surgery Clinic, Strängnäs (Other)
Responsible Party: Principal Investigator, Bo Nyström, Principal Investigator, Spinal Surgery Clinic, Strängnäs
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SpinalSC,SI
Record Dates: First submitted 2016-11-01; First posted 2016-11-11 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Pelvic Pain; Low Back Pain
MeSH Terms: conditions — Pelvic Pain; Low Back Pain | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgery (Experimental): Arthrodesis of SI-joint/s, physiotherapy
  Interventions: Procedure: Surgery
- Non-surgery (Active Comparator): Non-surgery, physiotherapy
  Interventions: Other: Non-surgery

INTERVENTIONS:
Procedure: Surgery — Arthrodesis of SI-joints, Physiotherapy
  Arms: Surgery
Other: Non-surgery — Physiotherapy
  Arms: Non-surgery

SUMMARY:
Background: Pelvic pain is common during pregnancy and usually subsides after delivery. Some women, however, experience severe and long-standing pelvic pain, judged to emanate from the Sacro-iliac joints (SI-joints). Radiological correlates are absent and there are diverging opinions regarding the value of different clinical testing procedures and the use of anaesthetic blocks to reveal SI-joint origin of the pain. In case of slight or moderate pain the situation may be solved by the use of analgetics and physical therapy, but in case of severe pain the situation might end up in a discussion whether surgery with arthrodesis of the SI joint might be of value. To our knowledge, however, the results from surgical treatment has not been compared with non-surgical treatment in a randomized study.

Aim: The investigators´ hypothesis is that

1. there exists a specific identifiable subgroup of patients within the chronic low back pain (CLBP) group in whom the pain emanates from the sacro-iliac (SI) joints, and that
2. patients in this subgroup may be selected based on thorough symptom analysis, and
3. that arthrodesis of the actual joint/s may reduce the pelvic pain. Methods: A RCT with parallel group design with pre- and post-treatment data. Inclusion of women 18-55 years old with pronounced pelvic pain for at least 2 years and having tried ordinary physical therapy without improvement and being on sick leave at least 50 percent. Operation by posterior approach with bone transplantation between the iliac bone and the sacrum, using microsurgical technique. Patients in both groups, the surgical (S) and non-surgical (NS) were all treated by formal physiotherapy at a five days stay at the Clinic and instructed to continue their training at home according to the lines given at the Clinic.

Outcome: The primary outcome was perceived pelvic pain according to the assessments on the validated Balanced Inventory for Spinal Disorders questionnaire (BIS) and on a Visual Analogue Scale (VAS) before treatment and at follow-up one year after treatment. The perceived change in pain was also assessed on a transitional scale in the follow-up version of the BIS.

Secondary patient reported outcome measures (PROM) were pain related functions assessed on the Oswestry Disability Index questionnaire (ODI), the BIS and the Roland-Morris questionnaire. Health related quality of life was assessed by using the Short-Form 36 (SF-36) and Euro-Quol (EQ-5D) questionnaires.

DETAILED DESCRIPTION:
Study description

1. a. Title Sacro-iliac joint arthrodesis or non-operative care for treatment of chronic pelvic pain.

   A randomized study.

   Introduction Background and objectives
2. a. Pelvic pain is common during pregnancy and usually subsides after delivery. Some women, however, experience severe and long-standing pelvic pain, judged to emanate from the SI-joints. Radiological correlates are absent and there are diverging opinions regarding the value of different clinical testing procedures and the use of anaesthetic blocks to reveal SI-joint origin of the pain. In case of slight or moderate pain the situation may be solved by the use of analgetics and physical therapy, but in case of severe pain the situation might end up in a discussion whether surgery with arthrodesis of the SI joint might be of value.

To our knowledge, however, the results from surgical treatment has not been compared with non-surgical treatment in a randomized study.

2 b. The investigators´ hypothesis is that

1. there exists a specific identifiable subgroup of patients within the chronic low back pain (CLBP) group in whom the pain emanates from the sacro-iliac (SI) joints, and that
2. patients in this subgroup may be selected based on thorough symptom analysis, and
3. that arthrodesis of the actual joint/s may reduce the pelvic pain.

   3 a. A RCT with parallel group design with pre- and post-treatment data. 3 b. No changes were made after trial commencement.

   Participant 4 a. Inclusion criteria Women 18-55 years old with pronounced pelvic pain for at least 2 years and having tried ordinary physical therapy without improvement and being on sick leave at least 50 percent.

   4 b. Eligible outpatients at the Clinic of Spinal Surgery, Strängnäs, Sweden, were informed about the study and those who consented to participate were included. The other women received ordinary treatment. Data were collected at the Clinic of Spinal Surgery, Strängnäs, Sweden.

   Interventions 5. A percutaneous mechanical provocation test was developed to obtain information regarding the possible pain origin in the SI joints. Injections with saline or local anaesthetics blind for the patients were performed against the posterior aspects of the SI joints, not intra-articular, to analyse the pain response at needle contact with the joint capsule, the pain reaction during injection and also the pain situation during the first hour after injection.

   Operation was performed by posterior approach with bone transplantation between the iliac bone and the sacrum, using microsurgical technique. Internal fixation was used.

   Patients in both groups, the surgical (S) and non-surgical (NS) were all treated by formal physiotherapy at a five days stay at the Clinic and instructed to continue their training at home according to the lines given at the Clinic.

   6 a. The primary outcome was perceived pelvic pain according to the assessments on the validated Balanced Inventory for Spinal Disorders questionnaire (BIS) and on a VAS before treatment and at follow-up one year after treatment. The perceived change in pain was also assessed on a transitional scale in the follow-up version of the BIS.

   Secondary patient reported outcome measures (PROM) were pain related functions assessed on the Oswestry Disability Index questionnaire (ODI), the BIS and the Roland-Morris questionnaire.

   Health related quality of life was assessed by using the SF-36 and EQ-5D questionnaires.

   6 b. No changes in the trial were made during the study.

   Sample size The sample size estimation was performed before study start by the statistician (ES). It was based on our previous experience of improvements in 55-60 % of the patients undergoing SI-joint arthrodesis compared to 10 % following physiotherapy. Assuming similar results of improvements a total sample size of 34 (17 + 17) will detect such a difference with the statistical power of 80 % (p < 0.05) when using statistical methods designed for change in rating scale assessments.

   7b. No interim analysis was performed.

   Randomization 8 a and b. A randomization scheme balanced for surgery /non-surgery patients was performed by using random permuted blocks in order to reduce predictability. A set of closed envelopes in numbered order with the message "operate" or "do not operate" was delivered to the Clinic by the statistician (ES) not involved in the treatment of the patients.

   Allocation concealment mechanism 9. The patients were consecutively included in the study according to the randomization envelopes.

   Implementation 10. A statistician not involved in the treatment of the patients generated the random allocation sequence. The surgeon enrolled the participants and a research nurse at the Clinic performed the practical assignment, i.e. opened the closed envelopes in consecutive order.

   Blinding 11 a. In accordance with the treatment alternatives the participants and the care givers could not be blinded to group assignment.

   11 b. Patients in both groups, the surgical and non-surgical, received equal treatment with formal physiotherapy. Besides, the patients in the surgical group were operated with arthrodesis.

   Statistical methods 12 a and b. The patients reported outcome variables (PROMs) were assessed on rating scales that generate ordered categorical data. Characteristic features are the ordered structure with lack of information regarding size and inter-categorical distances. Non-parametric rank-based statistical methods that take account of these limited mathematical properties of ordered categorical data are used for description and analysis. Frequency distribution, proportions, bar charts, median and quartiles are used for statistical descriptions. Statistical analysis of difference in outcomes assessed by transitional scales in the BIS by the two groups of patients was performed by the Wilcoxon-Mann-Whitney test. Statistical evaluation of change in the paired assessments made before treatment and on the follow-up occasion was made by Svensson´s methods for paired ordinal data that provides measures of systematic change in common for the group and additional measure of individual variability. The measures and the 95% confidence intervals of systematic change in position (RP), and in concentration (RC), and the measure of additional individual variability (RV) will be calculated as well as the differences in these measures between the two treatment groups. This statistical approach has been found to have a high power of detecting differences in small samples.

   Results 13. All patients in both groups received the allocated treatment and all patients in both groups were also seen at follow-up.

   Recruitment 14 a. Recruitment started October 22, 2008 and ended when the last patient was included in the study November 19, 2011.

   The follow-up took place from October 27, 2009 to November 19, 2012. 14 b. The trial was performed as planned but stopped after 3 years when 19 patients were included because of difficulties in recruiting eligible patients within reasonable time.

   16. The analyses will be carried out on the complete groups of 9 patients in the Surgery group and 10 patients in the NonSurgery group.

   17 a and b. The analyses are ongoing.

   Ancillary analysis 18. None.

   Harms 19. Will be reported when the analyses are completed.

   Comment Limitation 20. There was a small sample size because of difficulties in recruiting eligible patients, but a good research team and the choice of appropriate statistical analysis shows the power of this study.

   Generalizability 21. Provided that the patients being selected according to the same criteria as in the present study and the surgery being performed in the same way our results may be generalizable.

   22. During the last few years a remarkable increase is seen in the number of articles published concerning arthrodesis in case of presumed SI-joint pain, this due to the use of minimal invasive techniques. This increase in SI-joint surgery, however, is not a result of a better pre-operative evaluation of the patients. To our knowledge our study is the first RCT.

   Other information Registration 23. The study protocol was approved by the Regional Ethics Committee, Stockholm, (reference number 2008/289-31/3). In accordance with the Declaration of Helsinki, all patients were thoroughly informed concerning all parts of the study, both verbally and in written text, and gave their written informed consent.

   24. Then full trial protocol can be accessed via Bo Nyström, Clinic of Spinal Surgery, Strängnäs, Sweden, present address Regementsgatan 20 B, 64533 Strängnäs, Sweden.

   25. The study had no funding support.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18-55 years old with pronounced pelvic pain for at least 2 years.
2. Have tried ordinary physical therapy without improvement.
3. Being on sick leave at least 50 percent.

Exclusion Criteria:

Previous pelvic surgery.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2008-10; Primary Completion 2012-11 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Pelvic pain | One year
  Balanced Inventory for Spinal Disorders questionnaire
Pelvic pain | One year
  Visual Analogue Scale

SECONDARY OUTCOMES:
Function | One year
  ODI
Function | One year
  Roland-Morris Questionnaire

OTHER OUTCOMES:
Quality of life influenced by pelvic pain | One year
  SF-36, Low scores indicate a more impaired situation.
Quality of life influenced by pelvic pain | One year
  EQ-5D questionnaire, Low scores indicate a more impaired situation

IPD SHARING:
Plan to Share IPD: No